CLINICAL TRIAL: NCT07203261
Title: Comparison of the Body Roundness Index and A Body Shape Index With Body Fat and Visceral Fat in People Living With HIV: A Pilot Study
Brief Title: Comparison of the Body Roundness Index and A Body Shape Index With Body Fat and Visceral Fat in People Living With HIV.
Status: Not yet recruiting | Type: Observational
Sponsor: Queens College, The City University of New York (Other)
Responsible Party: Principal Investigator, Norberto Quiles, Associate Professor, Queens College, The City University of New York
Other Study IDs: TRADA-56-191
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: HIV/AIDS
Keywords: human immunodeficiency virus; Body composition
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV+: Participants living with HIV (HIV+) will have their waist circumference, hip circumference , height and weight measured. Participants will also have their body fat and visceral adipose tissue measured.

SUMMARY:
The study compares the Body Roundness Index (BRI) and the A Body Shape Index (ABSI) with with body fat and visceral fat in people living with HIV.

DETAILED DESCRIPTION:
Obesity is among the most prevalent cardiometabolic issues in recent years among people living with HIV (PLWH), and this is especially true among those that initiate and continue to take ART. Even newer first-line ART medications like Integrase inhibitors are strongly associated with the development of obesity among PLWH. This is of particular importance since research shows that excess fat, especially excess fat in the abdominal region, is associated with mortality (Jayedi et al., 2022; Lee et al., 2018). However, fat distribution in PLWH taking ART may not follow the same pattern of fat distribution found in general population (Lamesa et al., 2014). PLWH taking ART often experience abnormal accumulation of fat in the trunk and abdominal region (i.e., lipohypertrophy) and wasting of fat in the hips and extremities (i.e., lipoatrophy), both which can happen together or separately.

The Body Roundness Index (BRI) and A Body Shape Index (ABSI) are simple non- invasive anthropometric methods used to evaluate body fat distribution in general population. These measures can be very useful since they are predictive of overall body fat and visceral adipose tissue (VAT), and they correlate with diabetes, insulin resistance, metabolic syndrome among other cardiometabolic issues. Further, among PLWH, the ABSI and BRI have been associated with cardiovascular risk in men. However, the relationship between these anthropometric measures with overall body fat and VAT has not been evaluated among PLWH. The complex and unique nature of the fat distribution in PLWH taking ART warrants further evaluation of the validity of these measures in this patient population.

The study is cross-sectional in design and will be completed in one session. Participants living with HIV who agree to participate will be asked to complete a sociodemographic and health history questionnaire, and will then have their height, weight, waist circumference and hip circumference measured to calculate their BRI and ABSI. Participants will also have their body fat and lean body mass measured through air displacement plethysmography (ADP) and through bioelectrical impedance analysis (BIA). Visceral adiposity will be measured through ultra sound.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HIV
* Receiving the same anti-retroviral therapy for >= 6 months.

Exclusion Criteria:

* Pregnancy
* Having an implantable cardioverters or pacemakers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with HIV
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
A Body Shape Index | At enrollment, on the first day of the protocol.
  The ABSI is a measure of the body shape and the concentration of body volume. The ABSI is defined as the waist circumference (WC) divided by the body mass index (BMI) raised to two-thirds and by the square root of the person's height. WC will be measured just above the uppermost lateral border of the ilium at the end of a normal exhalation as recommended by NHANES guidelines. BMI will be calculated as Weight (kilograms) / Height (meters)2. Height will be measured using a standard stadiometer. With the participants without shoes. The measure will be taken with their back towards the stadiometer, buttocks touching the measurement surface, feet flat and externally rotated 60 degrees. The participants head will be aligned so that the horizontal line from the ear canal to the lower border of the orbit of the eye is parallel to the floor. The measure will be taken at the end of normal exhalation. Weight will be measured with the participant wearing minimal clothing and no shoes.
Body Roundness Index (BRI) | At enrollment, on the first day of the protocol.
  BRI is utilized to quantify the body shape of an individual using WC and height. WC will be measured just above the uppermost lateral border of the ilium at the end of a normal exhalation as recommended by NHANES guidelines. Height will be measured using a standard stadiometer. We will ask the participant to take off their shoes and stand with their back towards the stadiometer, with the buttocks touching the measurement surface at all times, feet flat and externally rotated approximately 60 degrees. Before taking the measurement we will align the participants head so that the horizontal line from the ear canal to the lower border of the orbit of the eye is parallel to the floor. The measure will be taken at the end of normal exhalation. Hip circumference will be measured at the widest part of the hip/buttocks area and will be added to increase the accuracy of the measure.
Visceral Adipose Tissue (VAT) | At enrollment, on the first day of the protocol.
  Visceral adipose tissue. VAT will be evaluated using the GE Logiq V2 ultrasound device. This measure will be used to evaluate the relationship between ABSI and BRI with VAT. The validity of ultrasound for measuring VAT has been established. The measurement will be taken using a 8 MHz abdominal probe transducer with the participant in supine position at the end of normal exhalation. Water based gel will be applied to the participants abdomen before the test. The transducer will be placed vertically against the skin in the saggital plane and pressed as lightly as possible to minimize the compression of the abdominal region. The distance between the posterior linea alba and the peritoneum immediately below, and 1 centimeter to the right of, the xiphoid process will be scanned. The measurement will be reported in centimeters.
Body fat (through bioelctrical impedance analysis; BIA) | At enrollment, on the first day of the protocol.
  Body fat will be measured using a Bioelectrical Impedance Analyzer (In body 770). The subject will stand on electrodes and grab a pair of electrodes. The test takes5 minutes and the analyzer is on for less than 1 minute. Body fat is calculated through the impedance or resistance of a low level electrical current passing through the body. Body fat percentage will be recorded.
Body fat (through air displacement plethysmography; ADP) | At enrollment, on the first day of the protocol.
  Body far will be measured through whole-body air displacement plethysmography (ADP) with estimated thoracic gas volume. Before the measurement we will ask the participant to change into a body forming swim suit and a swim cap. Then, we will ask the participant to sit inside the ADP chamber without moving for a couple of minutes while the equipment takes the measurements. The participant should not be able to feel anything while sitting inside the chamber. Thoracic gas volume will also be measured. Body density (D) is calculated from body mass (M) and measured body volume (V) using the formula: D = M / V. Body fat is calculated using the Siri equation: % Fat = (4.95 / D) - 4.5.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Physiology Laboratory, Flushing, New York, United States